CLINICAL TRIAL: NCT05630274
Title: A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LOXO-292 on the QTc Interval in Healthy Adult Subjects
Brief Title: A Study of Effect of Selpercatinib (LY3527723) on Corrected QT (QTc) Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17486; J2G-OX-JZJG (Other: Eli Lilly and Company); LOXO-RET-18032 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-11-21; First posted 2022-11-29 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: ABCD (Experimental): Period 1: 320 milligram (mg) Selpercatinib and Selpercatinib matching placebo (Treatment A) Period 2: 640 mg Selpercatinib (Treatment B) Period 3: 400 mg moxifloxacin (Treatment C) Period 4: Selpercatinib matching placebo (Treatment D) Participants received their assigned treatments in each of the above treatment period on Day 1 orally.
  Interventions: Drug: Selpercatinib
- Treatment Sequence 2: BDAC (Experimental): Period 1: 640 mg Selpercatinib (Treatment B) Period 2: Selpercatinib matching placebo (Treatment D) Period 3: 320 mg Selpercatinib and Selpercatinib matching placebo (Treatment A) Period 4: 400 mg moxifloxacin (Treatment C) Participants received their assigned treatments in each of the above treatment period on Day 1 orally.
  Interventions: Drug: Selpercatinib
- Treatment Sequence 3: CADB (Active Comparator): Period 1: 400 mg moxifloxacin (Treatment C) Period 2: Selpercatinib matching placebo (Treatment D) Period 3: 320 mg Selpercatinib and Selpercatinib matching placebo (Treatment A) Period 4: 640 mg Selpercatinib (Treatment B) Participants received their assigned treatments in each of the above treatment period on Day 1 orally.
  Period Title: Treatment Period 1
  Interventions: Drug: Moxifloxacin
- Treatment Sequence 4: DCBA (Placebo Comparator): Period 1: Selpercatinib matching placebo (Treatment D) Period 2: 400 mg moxifloxacin (Treatment C) Period 3: 640 mg Selpercatinib (Treatment B) Period 4: 320 mg Selpercatinib and Selpercatinib matching placebo (Treatment A) Participants received their assigned treatments in each of the above treatment period on Day 1 orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292
  Arms: Treatment Sequence 1: ABCD; Treatment Sequence 2: BDAC
Drug: Moxifloxacin — Administered orally
  Arms: Treatment Sequence 3: CADB
Drug: Placebo — Administered orally.
  Arms: Treatment Sequence 4: DCBA

SUMMARY:
The main purpose of this study is to assess the effect of Selpercatinib (LY3527723) on the heart rate-corrected QT (QTc) interval. The study will last up to 41 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, non-smoking, male or female (of non childbearing potential only or undergone sterilization procedures at least 6 months prior to the Screening) with no ECG abnormalities.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) at Screening and have a minimum weight of at least 50 kg at Screening
* Female of non childbearing potential: must have undergone sterilization procedures at least 6 months prior to the Screening
* Males who are capable of fathering a child must agree to use contraception from the time of the dose administration through 6 months after the last dose

Exclusion Criteria:

* Estimated creatinine clearance <90 milliliter per minute (mL/min) at Screening or Check in (Day -1; rechecks will be permitted up to two times to confirm participant eligibility for study participation).
* Has serum potassium levels <3.8 milliequivalents per liter (mEq/L) at Screening or Check in (Day -1; rechecks will be permitted up to two times to confirm participant eligibility for study participation).
* Has serum calcium levels < 8.5 milligrams/deciliter (mg/dL) at Screening or Check in (Day -1; rechecks will be permitted up to two times to confirm participant eligibility for study participation).
* Has serum magnesium levels <2.0 mEq/L at Screening or Check in (Day -1; rechecks will be permitted up to two times to confirm participant eligibility for study participation)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 4 treatment sequences (ABCD, BDAC, CADB, and DCBA), with each sequence having 4 periods where participants were crossed over between the periods. There was a washout period of 10 days between dosing in each period.
Groups:
- Treatment Sequence 3: CADB: Period 1: 400 mg moxifloxacin (Treatment C)
  Period 2: Selpercatinib matching placebo (Treatment D)
  Period 3: 320 mg Selpercatinib and Selpercatinib matching placebo (Treatment A)
  Period 4: 640 mg Selpercatinib (Treatment B)
  Participants received their assigned treatments in each of the above treatment period on Day 1 orally.
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: BDAC | Treatment Sequence 3: CADB | Treatment Sequence 4: DCBA
Started | 8 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: BDAC | Treatment Sequence 3: CADB | Treatment Sequence 4: DCBA
Started | 8 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: BDAC | Treatment Sequence 3: CADB | Treatment Sequence 4: DCBA
Started | 8 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: BDAC | Treatment Sequence 3: CADB | Treatment Sequence 4: DCBA
Started | 8 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Treatment Sequence 1: ABCD: Period 1: 320 mg Selpercatinib and Selpercatinib matching placebo (Treatment A)
  Period 2: 640 mg Selpercatinib (Treatment B)
  Period 3: 400 mg moxifloxacin (Treatment C)
  Period 4: Selpercatinib matching placebo (Treatment D)
  Participants received their assigned treatments in each of the above treatment period on Day 1 orally.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: BDAC | Treatment Sequence 3: CADB | Treatment Sequence 4: DCBA | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (11.44) | 40.3 (8.78) | 44.0 (8.88) | 10.18 (10.18) | 40.5 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 5 | 26
  Male | 1 | 0 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 4 | 4 | 14
  Not Hispanic or Latino | 6 | 4 | 4 | 4 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 5 | 6 | 6 | 8 | 25
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cardiodynamics: Placebo-corrected Change From Baseline in QT Interval Corrected Using Fridericia's Correction (QTcF) (ΔΔQTcF) for Treatments A, B, and C
Description: The cardiodynamic assessment was performed through 12-lead electrocardiogram (ECG) extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcF. Placebo-corrected change from baseline in QTcF (ΔΔQTcF) was calculated based on model-predicted effect
Time Frame: Pre-dose, -0.25, -0.5, -0.25, 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, and 24 hours post-dose
Population: All randomized participants who received at least one dose of selpercatinib or moxifloxacin with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- 320 mg Selpercatinib (Treatment A): Participants received single oral dose of 320 mg selpercatinib.
- 640 mg Selpercatnib (Treatment B): Participants received single oral dose of 640 mg selpercatinib.
- 400 mg Moxifloxacin (Treatment C): Participants received single oral dose of 400 mg moxifloxacin.
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B) | 400 mg Moxifloxacin (Treatment C)
Number analyzed (Participants) | 8 | 8 | 8
milliseconds | 3.4 [0.40 to 6.34] | 4.4 [1.37 to 7.40] | 6.4 [3.38 to 9.43]

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve From Time 0 to the Time of the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Description: PK: AUC0-t of Selpercatinib is reported.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, and 240 hours postdose
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per millilitre (ng*h/mL)
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
nanogram*hour per millilitre (ng*h/mL) | 33730 (42.3) | 42670 (65.8)

3. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib
Description: PK: AUC0-inf of Selpercatinib is reported.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
ng*hr/mL | 33830 (42.3) | 42830 (65.7)

4. Primary Outcome: PK: Percent of AUC0-inf Extrapolated (AUC%Extrap) of Selpercatinib
Description: PK: AUC%extrap of Selpercatinib is reported.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of AUC0-inf extrapolated
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
percentage of AUC0-inf extrapolated | 0.2986 (0.21464) | 0.3734 (0.53500)

5. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib is reported.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
nanogram per milliliter (ng/mL) | 2024 (74.6) | 2356 (103.0)

6. Primary Outcome: PK: Time to Reach Cmax (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib is reported.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
hour | 1.557 [0.80 to 24.06] | 2.051 [0.82 to 4.09]

7. Primary Outcome: PK: Apparent First Order Terminal Elimination Rate Constant (Kel) of Selpercatinib
Description: PK: Kel of Selpercatinib is reported.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
1/hour | 0.02515 (0.0087987) | 0.02459 (0.0070524)

8. Primary Outcome: PK: Apparent First-order Terminal Elimination Half-life (t½) of Selpercatinib
Description: PK: t½ of Selpercatinib is reported.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 320 mg Selpercatinib (Treatment A) | 640 mg Selpercatnib (Treatment B)
Number analyzed (Participants) | 32 | 31
hour | 31.189 (11.6988) | 30.582 (9.2791)

ADVERSE EVENTS:
Time Frame: Baseline up to 41 Days
Description: All participants who received at least one dose of the study drug. Per analysis plan adverse events were analyzed per each dose level.
Groups:
- 320 mg Selpercatinib: Participants received 320 mg Selpercatinib and administered orally on day 1.
- 640 mg Selpercatinib: Participants received 640 mg Selpercatinib administered orally on day 1.
- 400 mg Moxifloxacin: Participants received 400 mg moxifloxacin administered orally on day 1.
- Selpercatinib Matching Placebo: Participants received Selpercatinib matching placebo administered orally on day 1.
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 400 mg Moxifloxacin | Selpercatinib Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 6/32 | 2/32 | 0/32 | 4/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 320 mg Selpercatinib (N=32) | 640 mg Selpercatinib (N=32) | 400 mg Moxifloxacin (N=32) | Selpercatinib Matching Placebo (N=32)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT05630274/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT05630274/SAP_001.pdf